CLINICAL TRIAL: NCT04218396
Title: Evaluating the Efficacy and Feasibility of Virtual Reality Use for Peri-Procedural Analgesia and Anxiolysis: A Pilot Study
Brief Title: Virtual Reality Use for Peri-Procedural Analgesia and Anxiolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Linda Hung, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REB19-1907
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Acute Pain
Keywords: Acute Pain; Virtual Reality; Anxiolysis; Analgesia; Non-pharmacologic; Painful bedside procedure; Wound care; Dressing change
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment, Then Virtual Reality + Standard Treatment (Experimental): Participants will have an initial painful bedside procedure (eg: bedside wound care or dressing change) under standard treatment only. After a washout period, they then will have a repeat procedure (eg: similar bedside wound care or dressing change) under standard treatment AND virtual reality
  Interventions: Device: Virtual Reality use during painful bedside procedure; Drug: Standard Treatment during painful bedside procedure
- Virtual Reality + Standard Treatment, Then Standard Treatment (Experimental): Participants will have an initial painful bedside procedure (eg: bedside wound care or dressing change) under standard treatment AND virtual reality. After a washout period, they then will have a repeat procedure (eg: similar bedside wound care or dressing change) under standard treatment only.
  Interventions: Device: Virtual Reality use during painful bedside procedure; Drug: Standard Treatment during painful bedside procedure

INTERVENTIONS:
Device: Virtual Reality use during painful bedside procedure — Virtual reality (VR) will be used in addition to standard analgesic practices during painful bedside procedures. A head mounted display (HMD, Oculus Go Model #1KWPH812PN8354) and noise-cancelling headphones (Sony Model #MDRZ110B) will be provided to the patient during the procedure. This unit involves the patient wearing VR goggles, noise-cancelling headphones, and using a smartphone-based program with various applications the patient can choose from for analgesia/relaxation (eg: calming imagery/scenery of nature, activities involving mindfulness, interactive games or guided imagery, music and imagery, exercise imagery...etc). There are numerous, standard applications available for the patient to choose from, and the choice of most optimal application for analgesia, distraction, or anxiolysis will be left to the decision of the patient prior to their procedure.
Drug: Standard Treatment during painful bedside procedure — Pharmacologic sedation or high dose opioids (e.g. nurse-administered IV opioids, anxiolytics and sedatives, patient-controlled analgesia, anesthesiologist administered sedation, general anesthesia if required)

SUMMARY:
Currently, most analgesic regimens for painful bedside procedures rely on pharmacologic sedation or high doses of opioids (e.g.: nurse-administered IV opioids, anxiolytics, and sedatives; patient-controlled analgesia; anesthesiologist-administered sedation; and occasionally general anesthesia). Pharmacologic interventions are frequently associated with suboptimal analgesia, opioid-induced side effects, requirement for increased monitoring due to over sedation, and progressive acute tolerance to opioids over time, particularly with multiple/repeat procedures.

Alternative, non-pharmacologic strategies may help reduce pain, side-effects and opioid tolerance associated with painful bedside procedures. These strategies have not been studied as extensively, but are becoming more important in view of the current national opioid crisis. In particular, with recent technologic advancements, virtual reality (VR) has emerged as a non-pharmacologic modality for analgesia and anxiolysis, which can have tremendous benefits in acute pain management.

VR provides an immersive, realistic, often interactive experience for the user. It is frequently described as "transporting" the user to an alternate environment, with the use of high-fidelity head-mounted displays (HMD), noise-cancelling headsets, and a complete audio-visual experience. The user's sense of "presence" in the VR environment is crucial in providing patient engagement, and correlates with non-pharmacologic pain control.

VR has been shown to provide non-pharmacologic analgesia in children and adults undergoing painful procedures such as bedside wound care, burn treatment, and physical therapy. The use of VR during painful bedside procedures is one specific setting which offers a good starting point to investigate this technology for acute pain management.

Our study wishes to determine if VR plus standard therapy provides superior analgesia for painful bedside procedures (e.g. burn treatment, wound care) compared with standard therapy alone. Our primary outcome is a reduction in pain scores by 30%, as measured by a numerical analog scale (NAS) during painful bedside procedures. The investigators will use a randomized, cross-over study design in which hospitalized patients receiving repeated painful bedside procedures, will be randomized to 2 groups. Group A will have an initial painful bedside procedure under standard treatment only, and a repeat procedure under standard treatment + VR. Group B will have an initial procedure under standard treatment +VR, and a subsequent one under standard treatment. Questionnaires including pain scores and secondary outcomes will be administered to each patient before and after the bedside procedure. A convenience sample of patients will be recruited over 1 year (anticipated N~30).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing recurrent painful bedside procedures during hospitalization (at least 2 similar procedures during the course of hospital stay eg: wound dressing change)
* Anticipated duration of bedside procedure less than or equal to 2 hours
* Patients 18 years or older and able to provide informed consent
* Patients experiencing pain and/or anxiety from their bedside procedure (these patients are expected to benefit most from the analgesic/anxiolytic effects of VR).
* Patients who not wish to observe the painful bedside procedure (VR unit will provide sensory distraction and immersive experience, with HMD/goggles/headset, that allows patient not to witness procedure).
* Patients with adequate vision and hearing (with hearing aids if necessary) - patients with sensory limitations may not be able to benefit from the full effects of the VR sensory stimulation.
* Patients who are medically stable (should be free of acute conditions that could be dangerous when using VR)

Exclusion Criteria:

* Active seizure disorder, recent stroke (within 3 months), elevated intracranial pressure (visual and/or auditory stimulation may cause concerns with worsening acute central nervous system conditions)
* High risk for or active substance withdrawal; active substance intoxication (VR stimulation may worsen symptoms associated with substance intoxication and withdrawal)
* Active delirium (may preclude safe and effective use of VR as intended for anxiolysis and analgesia)
* Poor vision and hearing (precludes VR stimuli from being effective if the patient has sensory impairments that prevent them from seeing/hearing the VR effects)
* Open head/neck wound or head/neck injuries precluding safe use or wearing of the VR unit (headset, HMD, headphones)
* Body parasites, active eye infection, or other infectious diseases requiring contact isolation, droplet isolation, or airborne isolation (this exclusion limits the possibility of transmitting infectious diseases between patients with the use of the VR unit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-30 (Estimated); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-01-20 (Estimated)

PRIMARY OUTCOMES:
Numerical Analog Scale Pain Score | During painful bedside procedure
  The primary outcome is a reduction in pain scores by 30%, as measured by a numerical analog scale (NAS) during painful bedside procedures. Minimum scale value 0, maximum 10, higher scores mean more pain, lower scores mean less pain.

SECONDARY OUTCOMES:
Anxiety score - State Trait Anxiety Index short form questionnaire | During painful bedside procedure
  Anxiety score during painful bedside procedure as measured by State Trait Anxiety Index short form questionnaire. There are 6 separate statements ("I feel calm", "I am tense", "I feel upset", "I am relaxed", "I feel content", "I am worried"), minimum score on each question is 1, maximum score is 4. Lower scores indicate not feeling the emotion/state, and higher scores indicate feeling that emotion/state strongly.
Quality of life measures - Quality of Recovery 15 questionnaire | During painful bedside procedure
  Quality of Recovery 15 questionnaire - pain, nausea, psychometric data. Minimum score on first part of questionnaire (asking about positive features) is 0, maximum questionnaire score on first part of questionnaire is 100. On first part of questionnaire (asking about positive features), a lower score means a poorer outcome, a higher score means a better outcome. On the second part of the questionnaire, asking about negative experiences, the minimum score is 0, and the maximum score is 50. On the second part of the questionnaire (asking about negative features), a lower score means a better outcome, a higher score means a worse outcome.
Opioid use during painful bedside procedure | During painful bedside procedure
  Measurement of opioid use/requirement during painful bedside procedure (in morphine equivalents)
Number of participants with side effects related to virtual reality use during painful beside procedure (Nausea, dizziness, and other patient-reported adverse events) | During painful bedside procedure
  Nausea and other patient-reported adverse events side-effects and outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Linda Hung, MD, FRCPC, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Indovina P, Barone D, Gallo L, Chirico A, De Pietro G, Giordano A. Virtual Reality as a Distraction Intervention to Relieve Pain and Distress During Medical Procedures: A Comprehensive Literature Review. Clin J Pain. 2018 Sep;34(9):858-877. doi: 10.1097/AJP.0000000000000599. PMID 29485536
- [Background] Mallari B, Spaeth EK, Goh H, Boyd BS. Virtual reality as an analgesic for acute and chronic pain in adults: a systematic review and meta-analysis. J Pain Res. 2019 Jul 3;12:2053-2085. doi: 10.2147/JPR.S200498. eCollection 2019. PMID 31308733
- [Background] Gupta A, Scott K, Dukewich M. Innovative Technology Using Virtual Reality in the Treatment of Pain: Does It Reduce Pain via Distraction, or Is There More to It? Pain Med. 2018 Jan 1;19(1):151-159. doi: 10.1093/pm/pnx109. PMID 29025113